CLINICAL TRIAL: NCT05156567
Title: Multicenter Validation of a Multitask Deep Learning System for Spine Metastases Detection Andfeatures Evaluations at Spine Metastasis CT
Brief Title: Validation of a Multitask Deep Learning System at Spine Metastasis CT
Status: Completed | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhao Hui, Dr, Shanghai 6th People's Hospital
Other Study IDs: DLS01
Record Dates: First submitted 2021-12-12; First posted 2021-12-14 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: To Evaluate Performance of the DLS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- routine physicians
- DLS
  Interventions: Diagnostic Test: Deep Learning System

INTERVENTIONS:
Diagnostic Test: Deep Learning System — The multitask DLS with five algorithms detecting spine metastases and evaluate features (bone lesion quality, posterolateral involvement, and vertebral body collapse)
  Groups: DLS

SUMMARY:
15 resident oncologists were conducted to evaluate the clinical efficacy of DLS in multicenter. They were 1:1 randomly asked to independently read the test images without the assistance of DLS software or with the assistance. Area under the receiver operating characteristic curve (AUC), sensitivity, and specificity of the DLS were calculated with professional graders as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

1. pathology-proven diagnosis of solid tumor;
2. spinal CT scan indicating spinal metastasis with at least one lesion;
3. no previous surgery for spinal metastasis

Exclusion Criteria:

1. spinal CT scans with no sagittal reconstruction;
2. the radiologist considered that the quality of CT image was unqualified.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Spine Metastasis
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
AUC | 1 months
  Area under the receiver operating characteristic curve (AUC) of spinal instability detection

SECONDARY OUTCOMES:
sensitivity | 1 months
  sensitivity of spinal instability detection
specificity | 1 months
  specificity of spinal instability detection

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Sixth People's Hospital, Shanghai, China